CLINICAL TRIAL: NCT06567132
Title: Evaluation of the Effect of Non-Surgical Periodontal Treatment on IL-6, IL-10 and ANXA-1 Levels in Women With Polycystic Ovary Syndrome
Brief Title: Evaluation of the Effect of Non-Surgical Periodontal Treatment in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYASAR
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome; Gingivitis
Keywords: Annexin A1; Interleukin-6; Interleukin-10; Gingivitis; Polycystic ovary syndrome; Non-surgical periodontal treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Gingivitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Participants included in the study were divided into four groups according to whether they had polycystic ovary syndrome and gingivitis.
Who Masked: Outcomes Assessor
Masking Description: The person performing the biochemical analysis did not know the owner of the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PCOS and Healthy Periodontium (No Intervention): Women who are diagnosed with PCOS and have healthy periodontium. Clinical periodontal indices, saliva and gingival crevicular fluid samples were obtained.
- PCOS and Gingivitis (Active Comparator): Women who are diagnosed with PCOS and have gingivitis.Clinical periodontal indices, saliva and gingival crevicular fluid samples were obtained. Non-surgical periodontal treatment was performed.
  Interventions: Procedure: Non-surgical periodontal treatment
- Systemically healthy and Gingivitis (Active Comparator): Women who are systemically healthy and have gingivitis. Clinical periodontal indices, saliva and gingival crevicular fluid samples were obtained. Non-surgical periodontal treatment was performed.
  Interventions: Procedure: Non-surgical periodontal treatment
- Systemically and Periodontally Healthy (No Intervention): Women who are systemically healthy and have healthy periodontium. Clinical periodontal indices, saliva and gingival crevicular fluid samples were obtained.

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal treatment was performed in a single session using an ultrasonic device and a manual scaler. Polishing was done using polishing paste and rubber cup. Clinical periodontal indices, saliva and gingival crevicular samples were repeated after six weeks follow-up period.
  Other Names: Scaling and root planing
  Arms: PCOS and Gingivitis; Systemically healthy and Gingivitis

SUMMARY:
The goal of this clinical trial is to compare women with polycystic ovary syndrome and systemically healthy woman in relation to their gums and gum treatment outcomes as well as to investigate the role of a new biomarker in gum disease. The main questions it aims to answer are:

1. Is gum disease more common in women with PCOS?
2. Does PCOS affect the response to gum disease treatment?
3. Is there a new marker to identify gum disease? It is known that polycystic ovary syndrome is a low-grade chronic inflammatory disease. It has been reported that this aspect may be associated with gum disease. In our study, women with polycystic ovary syndrome will be compared with systemic healthy women. Initial gum conditions and response after treatment will be investigated. Additionally, the results will be supported by gingival crevicular fluid and saliva analysis.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine disorder characterized by hyperandrogenism, polycystic ovaries, and ovulatory dysfunction, affecting 4-21 % of women worldwide. It has been shown that PCOS has an impact on both local and systemic proinflammatory markers, along with periodontal disease, but the relationship between them remains unclear. The aim of this study is to compare the clinical and biochemical response to periodontal treatment between individuals with PCOS and gingival inflammation and those with systemic health, as well as to investigate the role of annexin-1 (ANXA1) biomarker in gingival inflammation.

Taking previous studies as a reference and considering the bleeding on probing variable as 45.12 and 82.94, respectively, and standard deviations as 37.46 and 13.59, respectively, the sample size for a 95% confidence level and 80% power at a 0.05 significance level was calculated as 15 people per group and n=60 in total. Considering that participants may drop out of the study, the sample size was determined as 20 people per group and n = 80 people in total.

A total of 80 participants were included, 40 individuals diagnosed with PCOS and 40 systemically healthy volunteers. Following periodontal examinations of all individuals, they were divided into four groups: a) PCOSPS (diagnosed with PCOS and healthy periodontium, n=20), b) PCOSG (diagnosed with PCOS and gingivitis, n=20), c) SG (systemically healthy individuals with gingivitis, n=20), and d) SPS (systemically healthy individuals with healthy periodontium, n=20). After gynecological and ultrasonographic examinations, as well as recording anthropometric measurements of all participants, hormonal tests were analysed. For the evaluation of periodontal status, clinical periodontal measurements were taken at the beginning of the study and at the 6th week after non-surgical periodontal treatment (NSPT) in the gingivitis groups. Gingival crevicular fluid (GCF) and saliva samples were collected at the beginning of the study and repeated at the 6th week after NSPT to assess the levels of interleukin-6 (IL-6), IL-10, and ANXA1. Biochemical analysis of all samples was performed using the enzyme-linked immunosorbent assay (ELISA) method.

An identification form was prepared to keep participants' records, including their personal and contact information. Gingival crevicular fluid tracking form to record when the gingival fluid samples were taken, which participant they belonged to, and from which dental area they were taken; saliva sample tracking form to record when the saliva samples were taken and which participant they belong to; periodontal index form to record plaque score, bleeding on probing, gingival pocket depth, gingival recession and attachment level during periodontal examination; polycystic ovary syndrome form containing the participants' medical information and a modified Ferriman-Gallwey score form was prepared to determine and record the degree of hirsutism.

Statistical analysis of the data obtained as a result of the study was performed in the IBM SPSS Statistics 26.0 program at a significance level of 0.05 and a confidence level of 95%. The distribution of the data was examined with the Shapiro-Wilk test. Comparisons between four independent groups with normal distribution were made with the One Way Anova test, and comparisons between four independent groups with non-normal distribution were made with the Kruskal Wallis test. Variables that were significant as a result of four group comparisons were compared with the Dunn-Bonferroni post-hoc test. If the variables met the assumption of normal distribution, comparisons between two independent groups were made with the Independent Sample t test. Chi-Square test or Fisher-Freeman-Halton test was used to evaluate the difference between categorical variables. In examining the relationship between numerical variables, Spearman (non-normally distributed) and Pearson (normally distributed) correlation coefficients were evaluated. The changes in time-dependent variables within and between groups were examined with the Repeated Anova test. While the descriptive statistics of the data were explained as mean and standard deviation or median (minimum-maximum), the descriptive statistics of categorical variables were given as frequency (%). ROC (Receiver Operating Characteristics) curve analysis was performed using Medcalc Version 12.3 to determine the distinctiveness of the ANXA1 variant.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 with polycystic ovary syndrome and healthy periodontium
* Women aged 18-40 with polycystic ovary syndrome and gingivitis
* Women aged 18-40 who are systemically healthy and have gingivitis
* Women aged 18-40 who are systemically healthy and have a healthy periodontium
* Presence of at least 20 permanent teeth

Exclusion Criteria:

* Receiving anti-inflammatory or antimicrobial therapy in the past three months
* Smoking and alcohol consumption
* Body mass index > 30 kg/m2
* Individuals with diabetes mellitus, hyperprolactinemia, congenital adrenal hyperplasia, androgen-secreting tumors, thyroid disorders, Cushing's syndrome, hypertension, liver or kidney dysfunction
* Medication that may affect metabolic criteria, such as oral contraceptive agents, any steroid hormone or related preparations, hypertensive drugs and insulin sensitizing drugs
* Pregnancy and breastfeeding
* Receiving periodontal treatment in the last 6 months
* Taking any medication known to affect periodontal status (e.g. phenytoin, calcium antagonists, cyclosporine, coumadin, steroidal non-anti-inflammatory drugs, aspirin > 81 mg)
* Active infectious diseases such as hepatitis, HIV or tuberculosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since polycystic ovary syndrome is a hormonal disorder seen in women, only female participants were eligible.
Enrollment: 80 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | Baseline and sixth weeks after the treatment
  Bleeding on probing is an important indicator of gingivitis. Bleeding on probing less than 10% is an indicator of healthy periodontium and means that the non-surgical periodontal treatment is successful.

SECONDARY OUTCOMES:
Interleukin-6 | Baseline and sixth weeks after the treatment
  Comparisons between groups were made by evaluating baseline and post-treatment levels.
Interleukin-10 | Baseline and sixth weeks after the treatment
  Comparisons between groups were made by evaluating baseline and post-treatment levels.
Annexin A1 | Baseline and sixth weeks after the treatment
  Comparisons between groups were made by evaluating baseline and post-treatment levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Assoc.Prof, Study Director — Affiliated; Cansu Can Yasar, Dr., Principal Investigator — Affiliated; Seda Ates, Prof., Study Chair — Affiliated
Locations (1):
- Bezmialem University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data could be shared if requested.

REFERENCES:
- [Background] Leite FRM, Nascimento GG, Moller HJ, Belibasakis GN, Bostanci N, Smith PC, Lopez R. Cytokine profiles and the dynamic of gingivitis development in humans. J Clin Periodontol. 2022 Jan;49(1):67-75. doi: 10.1111/jcpe.13565. Epub 2021 Oct 27. PMID 34664296
- [Background] Gonzalez F. Inflammation in Polycystic Ovary Syndrome: underpinning of insulin resistance and ovarian dysfunction. Steroids. 2012 Mar 10;77(4):300-5. doi: 10.1016/j.steroids.2011.12.003. Epub 2011 Dec 8. PMID 22178787
- [Background] Abraham Gnanadass S, Divakar Prabhu Y, Valsala Gopalakrishnan A. Association of metabolic and inflammatory markers with polycystic ovarian syndrome (PCOS): an update. Arch Gynecol Obstet. 2021 Mar;303(3):631-643. doi: 10.1007/s00404-020-05951-2. Epub 2021 Jan 13. PMID 33439300
- [Background] Bostanci N, Heywood W, Mills K, Parkar M, Nibali L, Donos N. Application of label-free absolute quantitative proteomics in human gingival crevicular fluid by LC/MS E (gingival exudatome). J Proteome Res. 2010 May 7;9(5):2191-9. doi: 10.1021/pr900941z. PMID 20205380
- [Result] Akcali A, Bostanci N, Ozcaka O, Gumus P, Ozturk-Ceyhan B, Tervahartiala T, Husu H, Buduneli N, Sorsa T, Belibasakis GN. Gingival Inflammation and Salivary or Serum Granulocyte-Secreted Enzymes in Patients With Polycystic Ovary Syndrome. J Periodontol. 2017 Nov;88(11):1145-1152. doi: 10.1902/jop.2017.170043. Epub 2017 Jun 9. PMID 28598286
- [Result] Akcali A, Bostanci N, Ozcaka O, Ozturk-Ceyhan B, Gumus P, Buduneli N, Belibasakis GN. Association between polycystic ovary syndrome, oral microbiota and systemic antibody responses. PLoS One. 2014 Sep 18;9(9):e108074. doi: 10.1371/journal.pone.0108074. eCollection 2014. PMID 25232962
- [Result] Akcali A, Bostanci N, Ozcaka O, Ozturk-Ceyhan B, Gumus P, Tervahartiala T, Husu H, Buduneli N, Sorsa T, Belibasakis GN. Elevated matrix metalloproteinase-8 in saliva and serum in polycystic ovary syndrome and association with gingival inflammation. Innate Immun. 2015 Aug;21(6):619-25. doi: 10.1177/1753425915572172. Epub 2015 Feb 23. PMID 25712810
- [Result] Ozcaka O, Buduneli N, Ceyhan BO, Akcali A, Hannah V, Nile C, Lappin DF. Is interleukin-17 involved in the interaction between polycystic ovary syndrome and gingival inflammation? J Periodontol. 2013 Dec;84(12):1827-37. doi: 10.1902/jop.2013.120483. Epub 2013 Jan 17. PMID 23327719
- [Result] Ozcaka O, Ceyhan BO, Akcali A, Bicakci N, Lappin DF, Buduneli N. Is there an interaction between polycystic ovary syndrome and gingival inflammation? J Periodontol. 2012 Dec;83(12):1529-37. doi: 10.1902/jop.2012.110588. Epub 2012 Apr 17. PMID 22509751
- [Result] Dursun E, Akalin FA, Guncu GN, Cinar N, Aksoy DY, Tozum TF, Kilinc K, Yildiz BO. Periodontal disease in polycystic ovary syndrome. Fertil Steril. 2011 Jan;95(1):320-3. doi: 10.1016/j.fertnstert.2010.07.1052. PMID 20800834
- [Result] Tarkun I, Cetinarslan B, Turemen E, Canturk Z, Biyikli M. Association between Circulating Tumor Necrosis Factor-Alpha, Interleukin-6, and Insulin Resistance in Normal-Weight Women with Polycystic Ovary Syndrome. Metab Syndr Relat Disord. 2006 Summer;4(2):122-8. doi: 10.1089/met.2006.4.122. PMID 18370758
- [Result] Casarin RCV, Salmon CR, Stolf CS, Paz HES, Rangel TP, Domingues RR, Pauletti BA, Paes-Leme AF, Araujo C, Santamaria MP, Ruiz KS, Monteiro MF. Salivary annexin A1: A candidate biomarker for periodontitis. J Clin Periodontol. 2023 Jul;50(7):942-951. doi: 10.1111/jcpe.13803. Epub 2023 Mar 19. PMID 36935103
- [Result] Hassan MN, Belibasakis GN, Gumus P, Ozturk VO, Emingil G, Bostanci N. Annexin-1 as a salivary biomarker for gingivitis during pregnancy. J Periodontol. 2018 Jul;89(7):875-882. doi: 10.1002/JPER.17-0557. PMID 29608211